CLINICAL TRIAL: NCT01931358
Title: Randomized, Double Blind Evaluation of Different One-Year Boosts After Sanofi Pasteur Live Recombinant ALVAC-HIV (vCP1521) and Global Solutions for Infectious Diseases (GSID) gp120 B/E (AIDSVAX® B/E) Prime-Boost Regimen in HIV-uninfected Thai Adults
Brief Title: Study of Boosting Strategies After Vaccination With ALVAC-HIV and AIDSVAX® B/E
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RV 306; WRAIR 1920 (Other: WRAIR IRB); S-11-0002 (Other: Sponsor)
Record Dates: First submitted 2013-08-12; First posted 2013-08-29 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX; AIDSVAX B-E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group Ia (Experimental): ALVAC-HIV at Weeks 0 and 4; ALVAC-HIV + AIDSVAX B/E at Weeks 12 and 24
  Interventions: Biological: ALVAC-HIV; Biological: AIDSVAX B/E
- Group Ib (Placebo Comparator): ALVAC-HIV Placebo at Weeks 0 and 4; ALVAC-HIV Placebo + AIDSVAX B/E Placebo at Weeks 12 and 24
  Interventions: Biological: ALVAC-HIV Placebo; Biological: AIDSVAX B/E Placebo
- Group IIa (Experimental): ALVAC-HIV at Weeks 0 and 4; ALVAC-HIV + AIDSVAX B/E at Weeks 12, 24 and 48
  Interventions: Biological: ALVAC-HIV; Biological: AIDSVAX B/E
- Group IIb (Placebo Comparator): ALVAC-HIV Placebo at Weeks 0 and 4; ALVAC-HIV Placebo + AIDSVAX B/E Placebo at Weeks 12, 24 and 48
  Interventions: Biological: ALVAC-HIV Placebo; Biological: AIDSVAX B/E Placebo
- Group IIIa (Experimental): ALVAC-HIV at Weeks 0 and 4; ALVAC-HIV + AIDSVAX B/E at Weeks 12 and 24; AIDSVAX B/E at Week 48
  Interventions: Biological: ALVAC-HIV; Biological: AIDSVAX B/E
- Group IIIb (Placebo Comparator): ALVAC-HIV Placebo at Weeks 0 and 4; ALVAC-HIV Placebo + AIDSVAX B/E Placebo at Weeks 12 and 24; AIDSVAX B/E Placebo at Week 48
  Interventions: Biological: ALVAC-HIV Placebo; Biological: AIDSVAX B/E Placebo
- Group IVa (Experimental): ALVAC-HIV at Weeks 0, 4 and 48; ALVAC-HIV + AIDSVAX B/E at Weeks 12 and 24
  Interventions: Biological: ALVAC-HIV; Biological: AIDSVAX B/E
- Group IVb (Placebo Comparator): ALVAC-HIV Placebo at Weeks 0, 4 and 48; ALVAC-HIV Placebo + AIDSVAX B/E Placebo at Weeks 12 and 24
  Interventions: Biological: ALVAC-HIV Placebo; Biological: AIDSVAX B/E Placebo

INTERVENTIONS:
Biological: ALVAC-HIV — 1 mL intramuscular injection containing 10^6 CCID50/dose
  Arms: Group IIIa; Group IIa; Group IVa; Group Ia
Biological: AIDSVAX B/E — 1 mL per injection (300 ug dose/antigen for a total of 600ug/dose administered)
  Arms: Group IIIa; Group IIa; Group IVa; Group Ia
Biological: ALVAC-HIV Placebo — 1 mL per injection
  Arms: Group IIIb; Group IIb; Group IVb; Group Ib
Biological: AIDSVAX B/E Placebo — 1 mL per injection
  Arms: Group IIIb; Group IIb; Group IVb; Group Ib

SUMMARY:
The primary purpose of the study is to better define the relative contributions of AIDSVAX® B/E alone, ALVAC-HIV alone, or ALVAC-HIV plus AIDSVAX® B/E combination to the observed immune profile in the weeks and months after receiving the original prime and boost vaccine regimen from study protocol RV 144, and their booster effects in both the systemic and mucosal compartments. In addition, this study will provide more intensive and comprehensive characterization of the innate, cell-mediated and humoral immune responses than possible within the RV 144 study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, HIV-uninfected male and female volunteers between age 20 and 40, weighing over 45 kilograms, and available for a period of 24 months and having a Thai identity card.
2. Must be at low risk for HIV infection per investigator assessment.
3. Must be able to understand and complete the informed consent process.
4. Must be capable of reading Thai.
5. Must successfully complete a Test of Understanding prior to enrollment.
6. Must be in good general health without clinically significant medical history.
7. HIV-uninfected per diagnostic algorithm within 45 days of enrollment.
8. Laboratory screening analysis:

   * Hemoglobin: Women ≥12.0 g/dL, Men ≥12.5 g/dL
   * White cell count: 4,000 to 11,000 cells/mm^3
   * Platelets: 150,000 to 450,000/mm^3
   * ALT and AST ≤1.25 institutional upper limit of reference range
   * Creatinine: ≤1.25 institutional upper limit of reference range
   * Urinalysis (dipstick) for blood and protein no greater than 1+ and negative glucose.
9. Female-Specific Criteria:

   * Negative pregnancy test for women at screening and prior to each vaccination(same day)and prior to any of the invasive procedures.
   * Be using adequate birth control methods for 45 days prior to the first vaccine/placebo vaccination and for at least 3 months after the final vaccine/placebo vaccination. Adequate birth control is defined as follows: Contraceptive medications delivered orally, intramuscularly, vaginally, or implanted, underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), condoms, diaphragms, intrauterine device (IUD), or abstinence.

Exclusion Criteria:

1. Asplenia: any condition resulting in the absence of a functional spleen.
2. Bleeding disorder diagnosed by a medical doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
3. Therapeutic anticoagulation resulting in an abnormal prothrombin (PT) / international normalized ration (INR) of partial prothrombin time (PTT).
4. Women breast-feeding or pregnant (positive pregnancy test) or planning to become pregnant during the window between study enrollment and 3 months after the last vaccination visit.
5. History of anaphylaxis or other serious adverse reaction to vaccines or allergies or reactions likely to be exacerbated by any component of the vaccine or placebo, including eggs, egg products, streptomycin, or neomycin.
6. Subject has received any of the following substances:

   * Chronic use of therapies that may modify immune response, such as IV immuneglobulin and systemic corticosteroids (in doses of > 20 mg/day prednisone equivalent for periods exceeding 10 days). The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least 2 weeks prior to enrollment in this study.
   * Blood products within 120 days prior to HIV screening.
   * Immunoglobulins within 30 days prior to HIV screening.
   * Any licensed vaccine within 14 days prior to initial study vaccine administration in the present study.
   * Receipt of any investigational HIV vaccine.
   * Investigational research agents or vaccine within 30 days prior to enrollment in the present study.
   * Anti-tuberculosis prophylaxis or therapy during the past 90 days prior to enrollment.
7. Active sexually transmitted infection confirmed by clinical exam and diagnostic test.
8. Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contradiction to protocol compliance or impairs a subject's ability to give informed consent.
9. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide ideation or attempt.
10. Study site employees who are involved in the protocol and/or may have direct access to study related area.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-09-24 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Immune Response | Through Week 96
  Characterization of vaccine-induced immune responses in the systemic and mucosal compartments by intracellular cytokine staining (ICS) and IFN-gamma ELISPOT at Baseline, Weeks 4, 12, 14, 24, 26, 36, 48, 50, 72 and 96.
Change in Humoral Immune Response | Through Week 96
  Characterization of vaccine-induced humoral immune response in the systemic and mucosal compartments by binding and neutralizing antibodies at Baseline, Weeks 4, 12, 14, 24, 26, 36, 48, 50, 72 and 96.

SECONDARY OUTCOMES:
Safety Monitoring | Through Week 48
  Post-vaccination reactions including erythema, induration, pain/tenderness, swelling and limitation of arm movement, fever, tiredness, chills, myalgia, arthralgia, headache, nausea, dizziness, and rash will be assessed and recorded on diary cards during the 3 days post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, MD, DTM&H, Principal Investigator — Mahidol University
Locations (3):
- Thailand (3):
  - Royal Thai Army Clinical Research Center, AFRIMS, Bangkok
  - Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok
  - Research Institute for Health Sciences (RIHES), Chiang Mai University, Chiang Mai

REFERENCES:
- [Background] Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Kaewkungwal J, Chiu J, Paris R, Premsri N, Namwat C, de Souza M, Adams E, Benenson M, Gurunathan S, Tartaglia J, McNeil JG, Francis DP, Stablein D, Birx DL, Chunsuttiwat S, Khamboonruang C, Thongcharoen P, Robb ML, Michael NL, Kunasol P, Kim JH; MOPH-TAVEG Investigators. Vaccination with ALVAC and AIDSVAX to prevent HIV-1 infection in Thailand. N Engl J Med. 2009 Dec 3;361(23):2209-20. doi: 10.1056/NEJMoa0908492. Epub 2009 Oct 20. PMID 19843557
- [Background] Rerks-Ngarm S, Paris RM, Chunsutthiwat S, Premsri N, Namwat C, Bowonwatanuwong C, Li SS, Kaewkungkal J, Trichavaroj R, Churikanont N, de Souza MS, Andrews C, Francis D, Adams E, Flores J, Gurunathan S, Tartaglia J, O'Connell RJ, Eamsila C, Nitayaphan S, Ngauy V, Thongcharoen P, Kunasol P, Michael NL, Robb ML, Gilbert PB, Kim JH. Extended evaluation of the virologic, immunologic, and clinical course of volunteers who acquired HIV-1 infection in a phase III vaccine trial of ALVAC-HIV and AIDSVAX B/E. J Infect Dis. 2013 Apr 15;207(8):1195-205. doi: 10.1093/infdis/jis478. Epub 2012 Jul 26. PMID 22837492
- [Derived] Shubin Z, Stanfield-Oakley S, Puangkaew J, Pitisutthithum P, Nitayaphan S, Gurunathan S, Sinangil F, Chariyalertsak S, Phanuphak N, Ake JA, O'Connell RJ, Vasan S, Akapirat S, Eller MA, Ferrari G, Paquin-Proulx D; for the RV306 Study Group. Additional boosting to the RV144 vaccine regimen increased Fc-mediated effector function magnitude but not durability. AIDS. 2023 Aug 1;37(10):1519-1524. doi: 10.1097/QAD.0000000000003611. Epub 2023 Jun 1. PMID 37260254
- [Derived] Pitisuttithum P, Nitayaphan S, Chariyalertsak S, Kaewkungwal J, Dawson P, Dhitavat J, Phonrat B, Akapirat S, Karasavvas N, Wieczorek L, Polonis V, Eller MA, Pegu P, Kim D, Schuetz A, Jongrakthaitae S, Zhou Y, Sinangil F, Phogat S, Diazgranados CA, Tartaglia J, Heger E, Smith K, Michael NL, Excler JL, Robb ML, Kim JH, O'Connell RJ, Vasan S; RV306 study group. Late boosting of the RV144 regimen with AIDSVAX B/E and ALVAC-HIV in HIV-uninfected Thai volunteers: a double-blind, randomised controlled trial. Lancet HIV. 2020 Apr;7(4):e238-e248. doi: 10.1016/S2352-3018(19)30406-0. Epub 2020 Feb 6. PMID 32035516